# **Statistical Analysis Plan**

# A Phase I, Open-label, Randomized, Parallel-arm, Single-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 133 Administered Subcutaneously in Healthy Japanese and Caucasian Subjects

SAP Status: Final SAP Version: 1.0 SAP Date: 18Nov2021

Investigational Medicinal Product: AMG 133

Protocol Reference: 20200290 Labcorp Study: 8473020

Sponsor: Amgen, Inc.

One Amgen Center Drive Thousand Oaks, California 91320

USA

Study Sites:

WCCT Global, LLC. 5630 Cerritos Avenue Cypress, California 90630

USA

Principal Investigators:

MD MPH MBE

Information described herein is confidential and may be disclosed only with the express written permission of the sponsor.

## TABLE OF CONTENTS

| TITLE PAGE | 1 |
|---|---|
| TABLE OF CONTENTS | 2 |
| LIST OF IN-TEXT TABLES AND FIGURES | 3 |
| LIST OF ABBREVIATIONS | 4 |
| 1. INTRODUCTION | 6 |
| 2. STUDY OBJECTIVES | 6 |
| 3. STUDY ENDPOINTS | 6 |
| 4. STUDY DESIGN | 7 |
| 5. SAMPLE SIZE JUSTIFICATION | 8 |
| 6. STUDY TREATMENTS | 8 |
| 7. DEFINITIONS OF POPULATIONS | 9 |
| 7.1. All Subjects Population | 9 |
| 7.2. Safety Population | 9 |
| 7.3. Pharmacokinetic Population | 9 |
| 8. STATISTICAL METHODOLOGY | 9 |
| 8.1. General | 9 |
| 8.1.1. Handling of Data Quality Issues Due to Coronavirus Disease 2019 and Re Restrictions | |
| 8.1.2. Calculation of the Summary Statistics | 10 |
| 8.1.3. Triplicate Readings | |
| 8.1.4. Repeat and Unscheduled Readings | 11 |
| 8.2. Subject Disposition and Population Assignment | 11 |
| 8.3. Screening Demographics and Baseline Characteristics | 12 |
| 8.4. Prior and Concomitant Medication | 12 |
| 8.5. Pharmacokinetic Assessments | 12 |
| 8.5.1. Pharmacokinetic Analysis | 12 |
| 8.5.2. Presentation of Pharmacokinetic Data | 14 |
| 8.5.3. Pharmacokinetic Statistical Methodology | 14 |
| 8.6. Safety and Tolerability Assessments | 15 |
| 8.6.1. Adverse Events | 15 |
| 8.6.2. Clinical Laboratory Parameters | 16 |

| 8.6.4. 12-lead Electrocardiogram Parameters | 17 |
|--------------------------------------------------------------|----|
| 8.6.5. Antibodies | 17 |
| 8.6.6. Other Assessments | 17 |
| 8.6.7. Safety and Tolerability Statistical Methodology | 17 |
| 9. INTERIM ANALYSES | 17 |
| 10. SIGNIFICANT CHANGES FROM THE PROTOCOL-SPECIFIED ANALYSES | 17 |
| 11. REFERENCES | 18 |
| 12. APPENDICES | 19 |
| Appendix 1: Document History | 19 |
| LIST OF IN-TEXT TABLES AND FIGURES | |
| Figure 1: Study Design | 8 |

## LIST OF ABBREVIATIONS

Abbreviations pertain to the statistical analysis plan (SAP) only (not the tables, figures, and listings [TFLs]).

%AUC<sub>extrap</sub> percentage of area under the plasma concentration-time curve due to

extrapolation from the last quantifiable concentration to infinity

ADaM Analysis Data Model

AE adverse event

AUC area under the concentration-time curve

AUC<sub>inf</sub> area under the plasma concentration-time curve from time zero

extrapolated to infinity

AUC<sub>last</sub> area under the plasma concentration-time curve from time zero to the

last quantifiable concentration

BLQ below the limit of quantification

CDISC Clinical Data Interchange Standards Consortium

CDER Center for Drug Evaluation and Research

CL/F apparent total clearance

C<sub>max</sub> maximum observed plasma concentration

COVID-19 coronavirus disease 2019
CRU clinical research unit
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

DMP data management plan
ECG electrocardiogram
EOS end of study

eCRF electronic case report form ICF informed consent form

ICH International Council for/Conference on Harmonisation

 $\lambda_z$  apparent terminal elimination rate constant

 $\lambda_z$  Lower start of exponential fit

 $\lambda_z$  N number of data points included in the log-linear regression  $\lambda_z$  Span Ratio time period over which  $\lambda_z$  was determined as a ratio of  $t_{1/2}$ 

 $\lambda_z$  Upper end of exponential fit

MedDRA Medical Dictionary for Regulatory Activities

NA not applicable PK pharmacokinetic(s)

R<sup>2</sup>-adj adjusted coefficient for determination of exponential fit

SAP statistical analysis plan

SC subcutaneous

SD standard deviation

SDV source document verification

 $t_{1/2}$  apparent terminal elimination half-life TEAE treatment-emergent adverse event

TFL table, figure, and listing

 $t_{last}$  time of the last quantifiable concentration

 $t_{max}$  time of the maximum observed plasma concentration  $V_z/F$  apparent volume of distribution during the terminal phase

WHODrug World Health Organization Drug Dictionary

## 1. INTRODUCTION

This SAP has been developed after review of the clinical study protocol (Amendment 1 dated 24 August 2021) and electronic case report form (eCRF).

This SAP describes the planned analysis of the pharmacokinetic (PK), safety, and tolerability data from this study. A detailed description of the planned TFLs to be presented in the clinical study report (CSR) is provided in the accompanying TFL shells document.

In general, the analyses are based on information from the protocol, unless they have been modified by agreement with Amgen Inc. A limited amount of information about this study (eg, objectives, study design) is given to help the reader's interpretation.

This SAP must be finalized prior to the lock of the clinical database. Additionally, the SAP and TFL shells should be finalized prior to any programming activities commencing.

This SAP supersedes any statistical considerations identified in the protocol; where considerations are substantially different, they will be so identified. If additional analyses are required to supplement the planned analyses described in this SAP, they may be performed and will be identified accordingly in the CSR. Any substantial deviations from this SAP will be agreed with Amgen Inc. and identified in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E3 guideline *Structure and Content of Clinical Study Reports*, ICH E8 guideline *General Considerations for Clinical Trials*, ICH E9 guideline *Statistical Principles for Clinical Trials*.<sup>1,2,3</sup>

The document history is presented in Appendix 1.

## 2. STUDY OBJECTIVES

The primary objective of the study is:

• to evaluate the PK of AMG 133 after single subcutaneous (SC) administration in healthy Japanese and Caucasian subjects.

The secondary objectives of the study are:

- to evaluate the safety and tolerability of AMG 133 after single SC administration in healthy Japanese and Caucasian subjects.
- to evaluate the incidence of anti-AMG 133 antibodies in healthy Japanese and Caucasian subjects.

#### 3. STUDY ENDPOINTS

The primary endpoints of the study are AMG 133 PK parameters:

• maximum observed plasma concentration (C<sub>max</sub>)

- area under the plasma concentration-time curve (AUC) from time zero to the last quantifiable concentration (AUC<sub>last</sub>)
- area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC<sub>inf</sub>).

The secondary endpoints of the study are:

- adverse events (AE)
- clinical laboratory tests
- 12-lead electrocardiograms (ECGs)
- vital signs
- incidence of anti-AMG 133 antibodies.

#### 4. STUDY DESIGN

This will be a Phase I, single-center, open-label, randomized, parallel-arm study to investigate the PK, safety, and tolerability of a single SC dose of AMG 133 in 3 groups of healthy Japanese subjects and 2 groups of healthy Caucasian subjects.

Approximately 35 subjects will be enrolled in total, with 7 subjects in each of the 5 groups.

Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to dose administration. Eligible subjects will be admitted into the clinical research unit (CRU) for Check-in on Day -1 and be confined to the CRU until clinic discharge on Day 8. On Day 1, 21 Japanese subjects will be randomly assigned in a 1:1:1 ratio to Group 1, 2, or 3, and 14 Caucasian subjects will be randomly assigned in a 1:1 ratio to either Group 4 or 5. Each subject will participate in 1 treatment group only.

On Day 1, AMG 133 will be administered as a single SC dose to the following groups:

• Group 1: mg (Japanese subjects)

• Group 2: mg (Japanese subjects)

• Group 3: mg (Japanese subjects)

• Group 4: mg (Caucasian subjects)

• Group 5: mg (Caucasian subjects)

The total duration of study participation for each subject (from Screening through end of study [EOS] visit) is anticipated to be approximately 21 weeks.

The start of the study is defined as the date the first enrolled subject signs an Informed Consent Form (ICF). The point of enrollment occurs at the time of subject number allocation.

The end of the study is defined as the date of the last subject's last assessment (scheduled or unscheduled).

An overview of the study design is shown in Figure 1.

Figure 1: Study Design



## 5. SAMPLE SIZE JUSTIFICATION

The sample size for this study is based practical considerations. No statistical hypotheses will be tested. Approximately 35 subjects will be enrolled across 5 groups (7 subjects per group). The study design and sample size per dose group for this study is considered adequate for evaluation of the study objectives.

## 6. STUDY TREATMENTS

The study treatment names, abbreviations, and ordering to be used in the TFLs are presented in Table.

Table 1:Presentation of Study Treatments in TFLs

| Treatments | | Abbreviation | | Order in TFLs |
|---|---|---|---|---|
| Group 1: | mg (Japanese subjects) | Japanese | mg AMG 133 | 1 |
| Group 2: | mg (Japanese subjects) | Japanese | mg AMG 133 | 2 |
| Group 3: | mg (Japanese subjects) | Japanese | mg AMG 133 | 3 |
| Group 4: mg (Caucasian subjects) | | Caucasian | mg AMG 133 | 4 |
| Group 5: | mg (Caucasian subjects) | Caucasian | mg AMG 133 | 5 |

All TFLs will be based on actual treatments (eg, if subject was assigned to receive Group 1 treatment but was wrongfully dosed with Group 3 treatment they would be summarized and listed under Group 3 treatment).


## 7. DEFINITIONS OF POPULATIONS

Any protocol deviations, including those due to coronavirus disease 2019 (COVID-19) and related restrictions (see Section 8.1.1), will be considered prior to database lock for their importance and taken into consideration when assigning subjects to populations.

## 7.1. All Subjects Population

The all subjects population will include all subjects who signed the ICF and had any study assessment recorded in the database per the protocol.

## 7.2. Safety Population

The safety population will include all subjects who received at least 1 dose of AMG 133.

## 7.3. Pharmacokinetic Population

The PK population will include all subjects who received at least 1 dose of AMG 133 and have evaluable PK data.

#### 8. STATISTICAL METHODOLOGY

#### 8.1. General

Listings will be provided for all data captured in the database, with the exception of medical history. Listings will include all subjects assigned to the all subjects population and include data up to the point of study completion or discontinuation. Subjects are generally considered to have completed the study if they complete the scheduled end of study visit (rather than early termination visit). Any subject who discontinues the study will be identified accordingly in the listings. Summaries and statistical analyses will include the subjects assigned to the relevant population based on data type.

Data analysis will be performed using the SAS® statistical software package Version 9.4 (or higher if a new version is issued during the study).

Analysis Data Model (ADaM) datasets will be prepared using Clinical Data Interchange Standards Consortium (CDISC) ADaM Version 2.1 (or higher if a new version is issued during the study) and CDISC ADaM Implementation Guide Version 1.2 (or higher if a new version is issued during the study). Pinnacle 21 Enterprise Version 4.2.0 (or higher if a new version is issued during the study) will be utilized to ensure compliance with CDISC standards.

Caution should be used when interpreting results from the statistical analyses conducted in this study because the sample size is not based on power calculations.

Where reference is made to 'valid' data, this refers to non-missing data which meet the predetermined criteria (eg, are not flagged for exclusion).

Where reference is made to 'all calculations', this includes, but is not limited to, summary statistics, statistical analyses, baseline derivation, changes from baseline, percentage changes from baseline, and any parameter derivations.

All figures will be produced on linear-linear or discrete-linear scales, as applicable, unless specifically stated otherwise.

# 8.1.1. Handling of Data Quality Issues Due to Coronavirus Disease 2019 and Related Restrictions

Due to COVID-19 and related restrictions, there is a high risk for impact to data integrity, with the recognized potential for:

- Missed visits, caused by, for example:
  - Subject unable to travel to site due to restrictions, the need to quarantine, or COVID-19 infection
  - o Subject unwilling to go to site due to fear of COVID-19 infection
  - Site postponing subject's visit due to investigator not being available (eg, if they have been dispatched to hospital handling COVID19 infections)
- Site unable to replenish supply of investigational product
- Incomplete data entry by sites due to limited resources to support study or no access to source documents or to eCRF
- Outstanding source document verification (SDV) due to sponsor or country restrictions on remote SDV, or no or limited access to site(s) for on-site visits
- Unanswered queries

At the time of the reporting of the study results, all protocol deviations due to COVID-19 or related restriction will be assessed for their severity and impact on the analyses. If needed, appropriate statistical methods will be applied as a mitigating action (eg, data might be categorized into 2 analysis groups, with and without COVID-19 and related restrictions impact); however, this will exclude any imputations of the missing values. Any mitigating actions will be agreed with Amgen Inc. in advance and identified in the CSR.

## 8.1.2. Calculation of the Summary Statistics

For continuous data the following rules will be applied:

- Missing values will not be imputed, unless specifically stated otherwise.
- Unrounded data will be used in the calculation of summary statistics.

• If the number of subjects with valid observations (n) <3, summary statistics will not be calculated, with the exception of n, minimum, and maximum.

• In general, as early termination data are not associated with any scheduled timepoint, they will be excluded from all calculations of summary statistics and statistical analyses. Exceptions may be made where justified.

For categorical data the following rules will be applied:

- For ordered categorical data (eg, AE severity), all categories between the possible minimum and maximum categories will be included, even if n = 0 for a given category.
- For non-ordered categorical data (eg, race), only those categories for which there is at least 1 subject represented will be included; unless specifically stated otherwise.
- Missing values will not be imputed, unless specifically stated otherwise. A 'missing' category will be included for any parameter for which information is missing. This will ensure that the population size totals are consistent across different parameters.

## 8.1.3. Triplicate Readings

For 12-lead electrocardiogram (ECG) data only, where triplicate readings are taken, the mean of triplicate readings will replace the separate individual triplicate readings in all calculations.

In case of incomplete triplicate readings (eg, only 2 out of 3 readings were recorded), the mean and/or medians will be calculated, as appropriate, based on the number of readings available.

## 8.1.4. Repeat and Unscheduled Readings

For vital signs and 12-lead ECG data only, any predose value recorded in addition to the original value or a postdose value recorded within 15 minutes of the original value will be defined as a repeat value; any postdose value recorded more than 15 minutes after the original value will be defined as an unscheduled value. For all other data types (eg, laboratory parameters), any value recorded in addition to the original value will be defined as an unscheduled value.

The original value will be replaced by the last associated repeat value in all calculations.

As unscheduled values are not associated with any scheduled timepoint, they will be excluded from all calculations.

## 8.2. Subject Disposition and Population Assignment

Subject disposition and population assignment will be listed.

A summary table by treatment will be provided, based on the safety population.

## 8.3. Screening Demographics and Baseline Characteristics

The screening demographics and baseline characteristics including sex, age, race, ethnicity, height, body weight, and body mass index will be listed.

A summary table by treatment will be provided, based on the safety population.

## 8.4. Prior and Concomitant Medication

Prior medication will be defined as medication that ends prior to dosing. Concomitant medication will be defined as medication that starts during or after dosing or starts but does not end prior to dosing.

Prior and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHODrug) Global, Format B3, Version September 2020 (or later if a new version is issued during the study; see the data management plan [DMP] for more details). Prior and concomitant medications will be listed.

#### 8.5. Pharmacokinetic Assessments

## 8.5.1. Pharmacokinetic Analysis

The following PK parameters will be determined where possible from the plasma concentrations of AMG 133 using noncompartmental methods in validated software program Phoenix WinNonlin (Certara, Version 8.1 or higher):

| Parameter | Units <sup>a</sup> | Definition |
|---|---|---|
| AUC <sub>last</sub> | h*μg/mL | area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration <sup>b</sup> |
| $\mathrm{AUC}_{\mathrm{inf}}$ | h*µg/mL | area under the plasma concentration-time curve from time zero extrapolated to infinity <sup>c</sup> |
| %AUC <sub>extrap</sub> | % | percentage of area under the plasma concentration-time curve<br>due to extrapolation from the last quantifiable concentration<br>to infinity |
| $C_{max}$ | $\mu g/mL$ | maximum observed plasma concentration |
| $t_{max}$ | h | time of the maximum observed plasma concentration |
| $t_{last}$ | h | time of the last quantifiable concentration |
| $t_{1/2}$ | h | apparent terminal elimination half-life |
| CL/F | L/h | apparent total clearance, calculated as Dose/AUCinf |
| $V_z/F$ | L | apparent volume of distribution during the terminal phase, |
| | | calculated as Dose/(AUC <sub>inf</sub> * $\lambda_z$ ) |

<sup>&</sup>lt;sup>a</sup> Units are based on concentration units (provided by the bioanalytical lab or preferred units for presentation of PK parameters) and dose units used in the study.

Additional PK parameters may be determined where appropriate.

<sup>&</sup>lt;sup>b</sup> The area under the concentration-time curve will be calculated using the linear trapezoidal (linear interpolation) rule.

<sup>&</sup>lt;sup>c</sup> Based on the last observed quantifiable concentration

Pharmacokinetic analysis will be carried out where possible using actual dose administered (mg) and actual postdose blood sampling times. If an actual time is missing, the sample concentration result will be treated as missing unless there is scientific justification to include the result using the nominal time.

The parameters C<sub>max</sub>, t<sub>last</sub>, and t<sub>max</sub> will be obtained directly from the concentration-time profiles. If C<sub>max</sub> occurs at more than 1 timepoint, t<sub>max</sub> will be assigned to the first occurrence of C<sub>max</sub>.

## 8.5.1.1. Criteria for the Calculation of Apparent Terminal Elimination Rate Constant and Half-life

The start of the terminal elimination phase for each subject will be defined by visual inspection and generally will be the first point at which there is no systematic deviation from the log-linear decline in concentrations.

The apparent terminal elimination rate constant ( $\lambda_z$ ) will only be calculated when a reliable estimate can be obtained using at least 3 data points, preferably not including C<sub>max</sub>, and the adjusted coefficient for determination of exponential fit ( $\mathbb{R}^2$ -adj) of the regression line is  $\geq 0.8$ . Parameters requiring  $\lambda_z$  for their calculation (eg, AUC<sub>inf</sub>, t<sub>1/2</sub>, CL/F, and V<sub>z</sub>/F) will only be calculated if the  $R^2$ -adj value of the regression line is  $\geq 0.8$ .

The following regression-related diagnostic PK parameters will be determined, when possible:

| Parameter | Units | Definition |
|---|---|---|
| $\lambda_{z}$ | 1/h | apparent terminal elimination rate constant |
| $\lambda_z$ Upper | h | end of exponential fit |
| $\lambda_z$ Lower | h | start of exponential fit |
| $\lambda_z N$ | NA | number of data points included in the log-linear regression |
| $\lambda_z$ Span Ratio | NA | time period over which $\lambda_z$ was determined as a ratio of $t_{1/2}$ |
| R <sup>2</sup> -adj | NA | adjusted coefficient for determination of exponential fit |

Where possible, the span of time used in the determination of  $\lambda_z$  (ie, the difference between  $\lambda_z$ Upper and  $\lambda_z$  Lower) should be  $\geq 2$  half-lives. If the  $\lambda_z$  Span Ratio is  $\leq 2$ , the robustness of the  $t_{1/2}$  values will be discussed in the CSR.

## 8.5.1.2. Criteria for Calculation and Reporting of Area Under the Concentration-time Curve

The minimum requirement for the calculation of AUC will be the inclusion of at least 3 consecutive concentrations above the lower limit of quantification. If there are only 3 consecutive concentrations, at least 1 should follow C<sub>max</sub>.

If the extrapolated area is >20%, AUC<sub>inf</sub> (and derived parameters, CL/F, and V<sub>z</sub>/F) may be excluded from the summary statistics and statistical analysis at the discretion of the sponsor or pharmacokineticist.


If AUC<sub>inf</sub> cannot be determined reliably for all subjects and/or dose levels, an alternative AUC measure, such as AUC to a fixed timepoint or AUC<sub>last</sub>, may be calculated.

# 8.5.1.3. Criteria for Handling Below the Limit of Quantification or Missing Concentrations for Pharmacokinetic Analysis

Plasma concentrations below the limit of quantification (BLQ) will be assigned a value of 0 before the first measurable concentration and thereafter BLQ concentrations will be treated as missing. The following rules apply to the specific situations defined below:

- If an entire concentration-time profile is BLQ, it will be excluded from PK analysis.
- Where 2 or more consecutive concentrations are BLQ at the end of a profile, the profile will be deemed to have terminated and any further quantifiable concentrations will be set to missing for the calculation of the PK parameters, unless they are considered to be a true characteristic of the profile of the drug.
- If a predose plasma concentration is missing, it will be set to 0 by default within Phoenix WinNonlin

## 8.5.1.4. Treatment of Outliers in Pharmacokinetic Analysis

If a value is considered to be anomalous due to being inconsistent with the expected PK profile, it may be appropriate to exclude the value from the PK analysis. However, the exclusion of any data must have strong justification and will be flagged in data listings and documented in the CSR.

Any quantifiable predose concentration value will be considered anomalous and set to missing for the PK analysis. This will be set to 0 by default in Phoenix WinNonlin.

#### 8.5.2. Presentation of Pharmacokinetic Data

If the actual time of sample collection deviates from the nominal time by more than  $\pm 20\%$ , the plasma concentration will be flagged and excluded from the summary statistics.

For plasma concentration data the following rules will apply:

- Values that are BLQ will be set to 0 for the calculation of summary statistics.
- Arithmetic mean or median values that are BLQ will be presented as 0.

For PK parameters the following rule will apply:

• Geometric mean and coefficient of variation will not be calculated for  $t_{last}$  or  $t_{max}$ .

## 8.5.3. Pharmacokinetic Statistical Methodology

All PK concentrations and parameters will be listed.

Summary tables, mean (+ standard deviation [SD]) figures, overlaying individual figures, and individual figures by treatment and time postdose will be provided for plasma PK concentrations. All figures will be produced on both linear and semi-logarithmic scales.

Summary tables by treatment will be provided for all PK parameters, with the exception of regression-related PK parameters.

## 8.6. Safety and Tolerability Assessments

#### 8.6.1. Adverse Events

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 24.0 (or higher if a new version is issued during the study; see the DMP for more details).

A treatment-emergent adverse event (TEAE) will be defined as an AE that starts during or after dosing, or starts prior to dosing and increases in severity after dosing.

A treatment-related TEAE will be defined as a TEAE with a relationship related to the study treatment, as determined by the investigator.

All AEs will be listed. In addition to the data recorded in the database, the listings will include derived onset time and duration. Onset time will be calculated from the time of dosing for TEAEs only.

The frequency of subjects with TEAEs and the number of TEAEs will be summarized for the following categories:

- TEAEs (overall, serious, leading to discontinuation, and leading to death) by treatment
- TEAEs by severity and treatment
- Treatment-related TEAEs (overall, serious, leading to discontinuation, and leading to death) by treatment
- Treatment-related TEAEs by severity and treatment

The frequency of subjects will be summarized separately for TEAEs and treatment-related TEAEs by the following:

- System organ class, preferred term, and treatment
- Preferred term and treatment

For the AE data the following rules will apply:

• For the derivation of treatment-emergent status (applicable to all AEs): If the start date/time of an AE is incomplete or missing, an AE will be assumed to not be a TEAE, unless the incomplete start date/time or the end date/time indicates an AE started after dosing.

- For the derivation of treatment-related status (applicable to TEAEs only): If the study treatment relationship for a TEAE is missing, a TEAE will be assumed to not be a treatment-related TEAE.
- For the derivation of onset time (applicable to TEAEs only): If the start date/time of a TEAE is missing, onset time will not be calculated. If the start date/time of a TEAE is incomplete, where possible, the minimum possible onset time will be calculated and presented in '≥DD:HH:MM' format (eg, if the date/time of dosing is 01MAY2019/08:00 and recorded start date/time of a TEAE is 03MAY2019, then the minimum possible onset time will be calculated by assuming a TEAE started at the first hour and minute of 03MAY2019 [03MAY2019/00:00], thus will be presented as onset time ≥01:16:00 in the listing). If the start date of a TEAE is the same as the date of dosing but the start time of a TEAE is missing, an onset time will be presented as '≥00:00:01'. Any clock changes will be accounted for in the derivation.
- For the derivation of duration (applicable to all AEs): If the end date/time of an AE is missing, duration will not be calculated. If the start or end date/time of an AE is incomplete, where possible, the maximum possible duration will be calculated and presented in '≤DD:HH:MM' format (eg, if the start of an AE date/time is 01MAY2019/08:00 and its recorded end date/time is 03MAY2019, then the maximum possible duration will be calculated by assuming an AE ended at the last hour and minute of 03MAY2019 [03MAY2019/23:59], thus will be presented as duration ≤02:15:59 in the listing). Any clock changes will be accounted for in the derivation.
- For the calculation of TEAE summary statistics: If the severity of a TEAE is missing, that TEAE will be counted under the 'missing' category.
- For the calculation of TEAE summary statistics: If a subject experienced multiple TEAEs with the same preferred term for the same treatment, this will be counted as 1 TEAE for that treatment under the maximum severity recorded.

## 8.6.2. Clinical Laboratory Parameters

All clinical laboratory parameters, will be listed, as applicable; any value outside the clinical reference range will be flagged. Separate listings will be provided for any parameter for which there is any individual subject value outside the respective clinical reference range.

Summary tables by treatment and timepoint will be provided for clinical chemistry and hematology parameters.

Values recorded as  $\langle x, \leq x, \rangle x$ , or  $\geq x$  will be displayed in the listings as recorded. For the derivation of listing flags, all calculations, and presentation in the figures, <x and <x values will be set to 0, whereas >x and  $\ge x$  values will be set to x.

#### 8.6.3. Vital Signs Parameters

All vital signs parameters will be listed, as applicable; any value outside the clinical reference range will be flagged.

Summary tables by treatment and timepoint will be provided by treatment group for all vital signs parameters as applicable.

## 8.6.4. 12-lead Electrocardiogram Parameters

All 12-lead ECG parameters will be listed; any value outside the clinical reference range will be flagged.

Summary tables by treatment and timepoint will be provided for all 12-lead ECG parameters.

#### 8.6.5. Antibodies

The formation of anti-AMG 133 antibodies will be summarized descriptively. The incidence and percentage of subjects who develop anti-AMG 133 antibodies (binding and if positive, neutralizing to native GLP-1) will be summarized by treatment group. Furthermore, the incidence and percentage of subjects with treatment boosted anti-AMG 133 antibodies will also be summarized. In addition, subjects with positive anti-AMG 133 binding antibody and anti-GLP-1 neutralizing antibody results will be listed individually with corresponding time points.

#### 8.6.6. Other Assessments

Medical history will not be listed.

All other safety and tolerability assessments not detailed in the above sections will be listed only.

## 8.6.7. Safety and Tolerability Statistical Methodology

No inferential statistical analyses are planned.

## 9. INTERIM ANALYSES

No interim analyses are planned.

## 10. SIGNIFICANT CHANGES FROM THE PROTOCOL-SPECIFIED ANALYSES

There were no significant changes from the protocol-specified analyses.


#### 11. REFERENCES

- 1. ICH. ICH Harmonised Tripartite Guideline: Structure and content of clinical study reports (E3). 30 November 1995.
- 2. ICH. ICH Harmonised Tripartite Guideline: General considerations for clinical trials (E8). 17 July 1997.
- 3. ICH. ICH Harmonised Tripartite Guideline: Statistical principles for clinical trials (E9). 5 February 1998.
- 4. Keene ON. The log transformation is special. Stat Med. 1995;14(8):811-819.
- 5. Brown H, Prescott R. Applied Mixed Models in Medicine. Chichester: John Wiley & Sons, 1999.
- 6. Statistical Approaches to Establishing Bioequivalence. Rockville, MD: US Dept of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER); January 2001.
- 7. Schuirmann DJ. A comparison of the two one sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987;15(6):657-680.

## 12. APPENDICES

# **Appendix 1: Document History**

| Status and Version | Date of Change | Summary/Reason for Changes |
|--------------------|----------------|----------------------------|
| Final Version 1.0 | NA | NA; the first version. |

NA = not applicable